CLINICAL TRIAL: NCT06534320
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Effects of Food in Single/Multiple Oral Administration of DA-302168S Tablets
Brief Title: Safety, Tolerability and Pharmacokinetic Characteristics Evaluation of DA-302168S Tablets
Acronym: DA168
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chendu DIAO Pharmaceutical Group CO., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-CP-DA168-01
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DA-302168S (Experimental): This study includes single-dose ascending and multiple-dose ascending studies. SAD study may contain 7 dose groups of 2.5 mg, 7.5 mg, 15 mg, 30mg, 50mg, 75mg and 100 mg. MAD study contains 1-4 dose groups which were evaluated in SAD study to be tolerated.
  Interventions: Drug: DA-302168S
- Placebo of DA-302168S (Placebo Comparator): This study includes single-dose ascending and multiple-dose ascending studies. SAD study may contain 7 dose groups of 2.5 mg, 7.5 mg, 15 mg, 30mg, 50mg, 75mg and 100 mg. MAD study contains 1-4 dose groups which were evaluated in SAD study to be tolerated.
  Interventions: Drug: Placebo of DA-302168S

INTERVENTIONS:
Drug: DA-302168S — SAD study may cotain 7 cohorts at dosage of 2.5 mg, 7.5 mg, 15 mg, 30 mg, 50 mg, 75 mg, 100 mg. Each cohort enrolls 6 subjects receive DA-302168S tablets.
  Arms: DA-302168S
Drug: Placebo of DA-302168S — SAD study may cotain 7 cohorts at dosage of 2.5 mg, 7.5 mg, 15 mg, 30 mg, 50 mg, 75 mg, 100 mg. Each cohort enrolls 2 subjects receive placebo of DA-302168S tablets.
  Arms: Placebo of DA-302168S
Drug: DA-302168S — MAD study may cotain 1-4 cohorts which were evaluated in SAD study to be tolerated . Each cohort enrolls 8 subjects receive study DA-302168S tablets.
  Arms: DA-302168S
Drug: Placebo of DA-302168S — MAD study may cotain 1-4 cohorts which were evaluated in SAD study to be tolerated . Each cohort enrolls 2 subjects receive study placebo of DA-302168S tablets.
  Arms: Placebo of DA-302168S

SUMMARY:
To Evaluate the Safety, Tolerability and Pharmacokinetics on DA-302168S Tablets in Randomized, Double-blind, Placebo-controlled Single-dose and Multiple-dose ascending Phase I Clinical Trials in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years old (including 18 and 55 years old), male or female.
* Weight: male ≥50kg, female ≥45kg, body mass index (BMI) in the range of 19.0 ~ 28.0kg/m2 (including the end value).
* Subjects and their spouses or partners did not plan to become pregnant or plan to donate sperm or ovum during the study period until 3 months after the last dose, and agreed to use at least one acceptable and effective contraceptive method.
* No clinically significant abnormalities identified in the judgement of investigator at screening.
* Written informed consent prior to any study specific procedures.

Exclusion Criteria:

* subjects with a history of abnormal clinical presentation, diseases to be excluded, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, endocrine system, renal, hepatic, gastrointestinal, respiratory, metabolic, and skeletal systems, and a history of malignant tumors, which are judged to be clinically significant by the Investigator.
* Use of any medication (including prescription, over-the-counter, herbal, etc.) or nutraceutical within 14 days prior to the first dose.
* May have any contraindications, allergies or hypersensitivity to DA-302168S Tablets (both test drug and placebo) or its excipients, GLP-1RA, DPP-4 analogues.
* Previous family history of medullary thyroid carcinoma or type 2 multiple endocrine adenoma syndrome.
* History or evidence of any of the following conditions:

  1. Decompensated heart failure (New York Heart Association (NYHA) Cardiac Classification III and IV [Appendix 5: NYHA Heart Failure Classification]), cardiac arrhythmias (e.g., supraventricular tachycardia, atrial fibrillation, atrial flutter, second or third degree atrioventricular block, QTcF intervals > 450 milliseconds for men or > 470 milliseconds for women [Appendix 8: Fridericia Method Corrected QT Interval Formula], PR intervals > 220 milliseconds, etc.) prior to the first administration of the study drug. (e.g., supraventricular tachycardia, atrial fibrillation, atrial flutter, grade II or III AV block, QTcF interval >450 ms in males or >470 ms in females [Appendix 8: Formula for Correcting QT Intervals by the Fridericia Method], PR interval >220 ms, etc.) and who, in the opinion of the investigator, are unsuitable for participation in this study;
  2. Serious trauma or acute infection that may affect glycemic control within 4 weeks prior to screening;
  3. Positive results for any of the Hepatitis B Surface Antigen, Hepatitis C Antibody, Syphilis Spirochete Antibody, or Human Immunodeficiency Virus (HIV) Antibody;
  4. Mental or neurological illness prior to screening, unwillingness to communicate, or a language barrier that prevents full understanding and cooperation;
  5. Other medical or psychiatric conditions that may increase the risk of participation in the study or that, in the judgment of the Investigator, may make the subject unsuitable for participation in the study, including a recent history (within the past two years) of major depression or other serious mental disorder, or any history of attempted suicide.
* Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg prior to the first dose and who, in the opinion of the investigator, are not suitable for participation in the study.
* Those who screen positive for substance abuse or have a history of substance abuse within the past five years or have used drugs in the 3 months prior to screening.
* Those who have participated in a clinical trial of another drug within 3 months prior to screening and have received any of the clinical trial drugs.
* Elective surgery was planned during the study period.
* Those who have donated or lost ≥200mL of blood, received a blood transfusion, or used blood products within 3 months prior to screening.
* Female subjects are pregnant or lactating.
* Those who consumed excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day, or who consumed tea, coffee and/or caffeinated beverages within 48 hours prior to the first dose of the drug, or who were unable to discontinue consumption during the trial period
* Previous chronic intake of xanthine- or grapefruit-rich beverages or foods, or consumption of any xanthine- or grapefruit-rich product within 48 hours prior to the first dose.
* Smokers or those who smoked an average of ≥5 cigarettes per day in the 3 months prior to screening, or those who were unable to stop using any tobacco-based products during the trial.
* Heavy drinkers or regular drinkers in the 3 months prior to screening, i.e., those who consume more than 14 standardized units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of 40% alcohol by volume spirits or 150 mL of wine) or those who have a positive breath test for alcohol at baseline or who are unable to discontinue the use of any alcohol-containing product during the test period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | SAD up to Day 5 and MAD up to Day 9.
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose in SAD phase. MAD study will be adjusted according to the SAD study.
  Plasma samples were collected at different points for pharmacokinetic analysis.
Tmax | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose in SAD phase. MAD study will be adjusted according to the SAD study.
  Plasma samples were collected at different points for pharmacokinetic analysis.
AUC0-t | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose in SAD phase. MAD study will be adjusted according to the SAD study.
  Plasma samples were collected at different points for pharmacokinetic analysis.
AUC0-∞ | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose in SAD phase. MAD study will be adjusted according to the SAD study.
  Plasma samples were collected at different points for pharmacokinetic analysis.
t1/2 | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose in SAD phase. MAD study will be adjusted according to the SAD study.
  Plasma samples were collected at different points for pharmacokinetic analysis.
CL/F | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose in SAD phase. MAD study will be adjusted according to the SAD study.
  Plasma samples were collected at different points for pharmacokinetic analysis.
Vd/F | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose in SAD phase. MAD study will be adjusted according to the SAD study.
  Plasma samples were collected at different points for pharmacokinetic analysis.
Kel | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose in SAD phase. MAD study will be adjusted according to the SAD study.
  Plasma samples were collected at different points for pharmacokinetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, Doctor, Principal Investigator — Gulou Hospital Affiliated to Nanjing Medical University
Locations (1):
- Gulou Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No